CLINICAL TRIAL: NCT03130972
Title: Etiology of Motor Developmental Delay in Children
Acronym: MDD
Status: Completed | Type: Observational
Sponsor: Bundang CHA Hospital (Other)
Responsible Party: Principal Investigator, MinYoung Kim, M.D., Professor, Bundang CHA Hospital
Other Study IDs: BD2015-129
Record Dates: First submitted 2016-11-15; First posted 2017-04-27 (Actual); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Delayed;Development;Physical; Delayed; Development, Intellectual

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- developmental delay: Children who visited tertiary rehabilitation clinic for delayed motor development were all included.

SUMMARY:
This study aims to identify the etiology of children with motor developmental delay, in association with the results of magnetic resonance imaging and genetic analysis.

DETAILED DESCRIPTION:
Results of other available assessments including Gross Motor Function Measurements and Bayley Scale of Infant Development, second edition, modified Ashworth Scale, IQ score and developmental language assessments are to be collected.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of motor developmental delay
* available results of functional assessments at ages older than 18 months Functional measures include either GMFM or BSID_II

Exclusion Criteria:

* single domain delay other than motor (e.g., speech delay)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children visiting tertiary hospital for motor developmental delay
Sampling Method: Non-Probability Sample
Enrollment: 1355 (Actual)
Dates: Start 2009-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change of Gross Motor Function Classification System from baseline at 6 months | through study completion, an average of 1 year
  To avoid variation in each individual the exact date of evaluation for every outcome is included to estimate the exact time from birth

SECONDARY OUTCOMES:
Brain MRI findings | From the date of the first documented developmental delay until the date of last documentation or date of death from any cause, whichever came first, assessed up to 100 months
  the first brain MRI taken after the event causative to developmental delay, read by radiology specialists
Mental quotient | From the date of the first documented developmental delay until the date of last documentation or date of death from any cause, whichever came first, assessed up to 100 months
  BSID-II mental month estimated/actual age in month times 100

IPD SHARING:
Plan to Share IPD: No